CLINICAL TRIAL: NCT01510743
Title: Incidence of Complication Depending on the Cannulation Site in US Guided Central Vein Catheterization
Brief Title: Ultrasound Guided Central Vein Catheterization and Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Assistant professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B1112_069_003
Record Dates: First submitted 2012-01-09; First posted 2012-01-16 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Brain Tumor
Keywords: open heart surgery; lung surgery; spine surgery; hepatobiliary surgery
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group SC (Active Comparator): US guided subclavian vein catheterization
  Interventions: Procedure: Catheterization of subclavian vein
- Group IJ (Active Comparator): US-guided internal jugular vein catheterization
  Interventions: Procedure: Catheterization of internal jugular vein

INTERVENTIONS:
Procedure: Catheterization of subclavian vein — Catheterization of subclavian vein
  Arms: Group SC
Procedure: Catheterization of internal jugular vein — Catheterization of internal jugular vein
  Arms: Group IJ

SUMMARY:
There has been no study comparing the complication rates between internal jugular vein catheterization and subclavian vein catheterization when they are performed using sonographic view. This prospective study would reveal the sort of complication and its rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgeries requiring central vein catheterizations for anesthetic management.

Exclusion Criteria:

* Refuse
* hematologic disorder
* Anatomical abnormalities of central vein structure

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1484 (Actual)
Dates: Start 2012-01-30 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
complication | during central vein catheterization and operation day
  any one of arterial puncture, hematoma, pneumothorax, hemothorax

SECONDARY OUTCOMES:
Access time | during central venous catheterization
  from penetration of skin to aspiration of venous blood into the syringe
Number of attempts | during central venous catheterization
  once/twice/three times
catheter tip placement | postoperative 1 day
  After reviewing the postoperative chest X ray film, we will check the position of the central venous catheter tip. The possible pisition of catheter tip is as follows:
  (1) Superior vena cava and Rirht Atrium junction (2)Right internal jugular vein (3)Left Internal jugular vein (4)Right Axillary vein (5)Lt. Axillary vein

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Hee Kim, Professor, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, Gyounggi, South Korea